CLINICAL TRIAL: NCT05704790
Title: Feasibility and Acceptability of Brief, Telehealth Cognitive Compensatory Training for Children Treated for Pediatric Cancer
Brief Title: Feasibility and Acceptability of Brief, Telehealth Cognitive Compensatory Training for Pediatric Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UMCC 2022.068; HUM00218780 (Other: University of Michigan)
Record Dates: First submitted 2023-01-09; First posted 2023-01-30 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Pediatric Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): The intervention will include 5 weekly sessions (60-90 minutes each) of cognitive compensatory training (CCT) delivered virtually by a pediatric neuropsychologist.
  Interventions: Other: Cognitive Compensatory Training

INTERVENTIONS:
Other: Cognitive Compensatory Training — The intervention will include 5 weekly sessions (60-90 minutes each) of cognitive compensatory training (CCT) delivered virtually by a pediatric neuropsychologist.

SUMMARY:
This pilot study will be a prospective, single arm study to investigate the feasibility and acceptability of a brief, telehealth, cognitive compensatory training intervention for children with a history of pediatric cancer at the University of Michigan. Study aims to enroll 10 children with a history of treatment for pediatric cancer, along with their caregiver.

ELIGIBILITY:
Inclusion Criteria:

* Patient between the ages of 8 and 18
* Patient has a history of pediatric cancer
* Patient is at least 6 months posttreatment completion
* Patient and caregiver are fluent in English, as intervention materials are only available in English at this time.
* Patient demonstrates deficits in attention and/or executive functioning as evidenced by either (a) performance below one standard deviation on at least one cognitive measure of attention or executive functioning, such as on the Conners Continuous Performance Test (CPT-3), Trail making Test A & B, Children's Category Test (CCT), and Wisconsin Card Sorting Test (WCST) and/or (b) executive functioning and attention problems are identified during screening with the research assistant.

Exclusion Criteria:

* Patient has a history of treatment for a pediatric brain tumor
* Patient has a history of traumatic brain injury or seizures
* Patient has a history of a developmental disorder (i.e., autism, intellectual disability), behavioral disorder (i.e., oppositional defiant disorder, conduct disorder), or mood disorder (i.e., disruptive mood dysregulation disorder) that would negatively interfere with patient's participation in the intervention.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2023-02-17 (Actual); Primary Completion 2024-07-23 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
Determining satisfaction and perceived benefit from study intervention based off of change in results from the BRIEF-2 questionnaire from baseline to 6 weeks post trial entry | 6 weeks from trial entry
  Completion of Study Questionnaire, BRIEF-2, at time of enrollment at after intervention completion.
Determining satisfaction and perceived benefit from study intervention based off of change in results from the Conners 3 questionnaire from baseline to 6 weeks post trial entry | 6 weeks from trial entry
  Completion of Study Questionnaire, Conners 3, at time of enrollment at after intervention completion.
Determining satisfaction and perceived benefit from study intervention based off of change in results from the SMALSI-2 questionnaire from baseline to 6 weeks post trial entry | 6 weeks from trial entry
  Completion of Study Questionnaire, SMALSI-2, at time of enrollment at after intervention completion.
Determining satisfaction and perceived benefit from study intervention based off of change in results from the SPSI-R questionnaire from baseline to 6 weeks post trial entry | 6 weeks from trial entry
  Completion of Study Questionnaires, SPSI-R , at time of enrollment at after intervention completion.
Determining satisfaction and perceived benefit from study intervention based off of change in results from the PKEQ questionnaire from baseline to 6 weeks post trial entry | 6 weeks from trial entry
  Completion of Study Questionnaires, PKEQ, at time of enrollment at after intervention completion.

OTHER OUTCOMES:
Study completion | 6 weeks from trial entry
  Possible factors contributing to study completion will be gathered from the History Questionnaire
Clinical outcomes based off of response to the BRIEF-2 study questionnaire | 6 weeks from trial entry
  Clinical outcomes of the intervention will also be summarized using empirically validated caregiver and child responses to the BRIEF-2 questionnaire
Clinical outcomes based off of response to the Conners 3 study questionnaire | 6 weeks from trial entry
  Clinical outcomes of the intervention will also be summarized using empirically validated caregiver and child responses to the Conners 3 questionnaire
Clinical outcomes based off of response to the SMALSI-2 study questionnaire | 6 weeks from trial entry
  Clinical outcomes of the intervention will also be summarized using empirically validated caregiver and child responses to the SMALSI-2 questionnaire
Clinical outcomes based off of response to the SPSI-R study questionnaire | 6 weeks from trial entry
  Clinical outcomes of the intervention will also be summarized using empirically validated caregiver and child responses to the SPSI-R questionnaire
Clinical outcomes based off of response to the PKEQ study questionnaire | 6 weeks from trial entry
  Clinical outcomes of the intervention will also be summarized using empirically validated caregiver and child responses to the PKEQ questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Kaitlin McCloskey, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
PI does not plan to share IPD